CLINICAL TRIAL: NCT07050511
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Sequential Group, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GB-0669 in Healthy Subjects
Brief Title: Study to Investigate the Safety, Tolerability, and Pharmacokinetics of GB-0669 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Generate Biomedicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GB-0669-101
Record Dates: First submitted 2025-05-21; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: SARS CoV-2
Keywords: SARS CoV-2; GB-0669

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Intervention GB-0669 (Experimental): Study intervention
  Interventions: Drug: GB-0669
- Placebo (Placebo Comparator): sterile 0.9% (w/v) sodium chloride solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GB-0669 — Single IV infusion of GB-0669.
  Arms: Study Intervention GB-0669
Drug: Placebo — Single IV infusion of placebo. Sterile 0.9% (w/v) sodium chloride solution.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test the safety and tolerability of a single ascending dose (SAD) of GB-0669 administered intravenously in adults. The goal of this study is also to measure the blood levels of GB-0669 in the body.

Study participants will be assigned to receive the study drug or placebo (the placebo is called saline; it is a liquid like salt water and made to look like the study drug but contains no active ingredient).

The study is blinded, which means you and the study doctor will not know whether you are getting the study drug or placebo.

Study participants will be assigned to one of 5 cohorts (study groups). Each cohort will have a single ascending dose (SAD). The first two SAD cohorts will have 3 study participants receiving GB-0669 and 3 study participants receiving placebo. The last three SAD cohorts will have 10 study participants receiving GB-0669 and 3 study participants receiving placebo. The SAD cohort dose levels will be as follows: 100 mg, 300 mg, 600 mg, 1200 mg, 2400 mg.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled first in human (FIH) trial to evaluate the safety, tolerability, and pharmacokinetics of GB-0669 in healthy study participants. The trial is designed to administer the GB-0669 drug product intravenously at 5 single ascending dose (SAD) cohort dose levels.

Eligible study participants will be screened and randomized to receive either GB-0669 or placebo in each cohort. The safety of the participants enrolled in this trial will be carefully monitored. There will be an independent safety review committee (iSRC) that will review ongoing safety for this trial and provide recommendations to proceed with the cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects
2. Adults, 18 to 55 years of age (inclusive) at screening
3. Body mass index (BMI) ≥ 19.0 and ≤ 35.0 kg/m2
4. Medically healthy without clinically significant abnormalities at screening and pre-dose on Day 1
5. Negative SARS-CoV-2 rapid antigen or PCR tests prior to randomization
6. Physical examination without any clinically relevant findings
7. Systolic blood pressure in the range of 90 to 140 mmHg and diastolic blood pressure in the range of 50 to 90 mmHg after 5 minutes in seated, semi-recumbent, or supine position
8. Heart rate (HR) in the range of 50 to 100 bpm after 5 minutes rest in seated, semi-recumbent, or supine position
9. Body temperature, between 35.0°C and 37.5°C
10. In the opinion of the investigator, no significant findings in serum chemistry, hematology, coagulation, and urinalysis tests
11. Female subjects of childbearing potential, defined as any woman who has experienced menarche and who is not permanently sterile or postmenopausal, must have negative blood pregnancy tests at screening (and negative urine pregnancy tests on Day 1) and must agree to use protocol-defined methods of contraception from screening through at least 90 days after study completion
12. Male subjects must agree to use protocol-defined methods of contraception and agree to refrain from donating semen from screening through at least 90 days after study completion
13. Have suitable venous access for intravenous infusion and blood sampling
14. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions including staying overnight in the CRU.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, oncological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease, including any acute illness or surgery within the past 3 months determined by the principal investigator (PI) to be clinically relevant. Subjects with localized cancers treated with curative intent and not on active therapy are allowed
2. Current infection that requires antibiotic, antifungal, antiparasitic or antiviral medications
3. Acute illness or fever within 3 days before study enrollment (enrollment may be delayed for full recovery if acceptable to the investigator)
4. Abnormal EKG or any known cardiac condition determined by the PI to be clinically Current infection that requires antibiotic, antifungal, antiparasitic or antiviral medications
5. Positive testing for any of the following: human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C antibodies (HCV)
6. Women currently pregnant, lactating, or planning a pregnancy between enrollment and final study visit, or intends to donate ova during this time period
7. Male participants intend to donate sperm during this study or before the end of the study
8. Any history of anaphylactic-type reaction to any substance or any history of infusion related reactions or any allergy to components of the study drug
9. Blood donation or significant blood loss (i.e., > 500 mL) within 56 days prior to Day 1
10. Plasma donation within 7 days prior to Day 1
11. Use of more than an average of 5 packs/week of tobacco/nicotine-containing product within 6 months prior to Day 1. Subjects must agree to refrain from smoking for the duration of the study
12. Excessive intake of alcohol, defined as an average daily intake of greater than 2 standard drinks for women and 4 standard drinks for men, (1 bottle of beer (375mL) is equivalent to approximately 1.4 standard drinks, 1 glass of spirits (30mL) is equivalent to approximately 1 standard drink and 1 glass (150mL) of wine is equivalent to approximately 1.5 standard drinks)
13. History of alcohol abuse, illicit drug use, physical dependence to any opioid, or any history of drug abuse or addiction within 2 years prior screening
14. Individuals currently participating or planning to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, or medication); or who have received an experimental agent within 1 month (or 3 half-lives) before enrollment of this study; or expect to receive another experimental agent during participation of this study
15. Positive urine test for drugs of abuse or alcohol (legal amounts of tetrahydrocannabinol (THC) are allowed)
16. Unwilling or unlikely to comply with the requirements of this study
17. Any condition or disease that, in the opinion of the Investigator, would pose a risk to participant safety or interfere with study evaluation, procedures or completion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 51 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of a single ascending dose of GB-0669 administered intravenously in healthy volunteers | Day -1 to Day 302
  Participant incidence and severity of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and TEAEs leading to discontinuation of study treatment. Clinically significant (CS) changes from baseline in: Clinical laboratory results (hematology, clinical chemistry, coagulation and urinalysis, vital signs, twelve-lead electrocardiograms (ECGs).

SECONDARY OUTCOMES:
To characterize the maximum concentration (Cmax) of GB-0669 following single doses of GB-0669 administered intravenously in healthy volunteers | Day 1 to Day 302
  The Cmax of GB-0669 following single doses in healthy volunteers will be analyzed
To characterize the time to peak drug concentration (Tmax) of GB-0669 following single doses of GB-0669 administered intravenously in healthy volunteers | Day 1 to Day 302
  The Tmax of GB-0669 following single doses in healthy volunteers will be analyzed
To characterize the half-life (t1/2) of GB-0669 following single doses of GB-0669 administered intravenously in healthy volunteers | Day 1 to Day 302
  The t1/2 of GB-0669 following single doses in healthy volunteers will be analyzed
To characterize the area under the curve to last quantifiable timepoint (AUClast) of GB-0669 following single doses of GB-0669 administered intravenously in healthy volunteers | Day 1 to Day 302
  The AUClast of GB-0669 following single doses in healthy volunteers will be analyzed
To characterize the volume of distribution (V/F) of GB-0669 following single doses of GB-0669 administered intravenously in healthy volunteers | Day 1 to Day 302
  The V/F of GB-0669 following single doses in healthy volunteers will be analyzed
To characterize the area under the plasma concentration- time curve (AUC) of GB-0669 following single doses of GB-0669 administered intravenously in healthy volunteers | Day 1 to Day 302
  The AUC of GB-0669 following single doses in healthy volunteers will be analyzed
To characterize the total body clearance from plasma (CL/F) of GB-0669 following single doses of GB-0669 administered intravenously in healthy volunteers | Day 1 to Day 302
  The CL/F of GB-0669 following single doses in healthy volunteers will be analyzed
To characterize the area under the plasma concentration-time curve from time zero to infinity (AUCinf) of GB-0669 following single doses of GB-0669 administered intravenously in healthy volunteers | Day 1 to Day 302
  The AUCinf of GB-0669 following single doses in healthy volunteers will be analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Generate Biomedicines, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This study was a Phase 1 trial conducted in healthy volunteers to assess safety and pharmacokinetics. Individual participant data will not be shared due to the limited clinical relevance of the data outside the context of internal decision-making and the absence of participant consent for external data sharing. The data are being used to support ongoing product development and regulatory interactions.